CLINICAL TRIAL: NCT06817317
Title: The Effect of Two Different Learning Methods on the Perception of Disaster Preparedness and Competences Related to Disaster Management in Nursing Students: a Randomized Controlled Trial
Brief Title: The Effect of Two Different Learning Methods on Disaster Perception and Management in Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Enise Sürücü, Dr., Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/08
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Students, Nursing; Learning Techniques
Keywords: peer education; self learning; model based training; disaster preparedness; disaster management

STUDY DESIGN:
Intervention Model Description: Intervention group: Model Based Training Group; Intervention group: Peer and Self-Learning Group; Control group: routine education programme
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Group 1 (Experimental): In this study, 'Disaster Nursing' course is an elective course integrated into the nursing curriculum. Disaster nursing course content to be applied to the Model based training group; the topics related to pre-disaster, disaster, post-disaster and recovery phases were prepared in line with International Nurses Association (ICN) Basic Competence Areas in Disaster Nursing, General Directorate of Emergency Health Services First Aid Training Guide and Jenning's Disaster Management Model in Nursing.
  One day a week for 5 weeks, the theoretical part 100 minutes (transferred by the academic staff responsible for the course), laboratory 50 minutes (transferred by theNational Medical Rescue Team personnel).
  There are 20 students in this group. Data were collected through data collection tools at pre-intervention, 5-week post-intervention, 1st month follow-up, 3rd month follow-up and 6th month follow-up stages.
  Interventions: Other: Model Based Training
- Intervention Group 2 (Experimental): In this study, peer and self-learning group consisted of four different seminar groups of five students randomised. The students were informed about creating a seminar programme on disaster nursing and management and making presentations until the dates determined at the beginning of the semester. It was explained that they would use peer and self-learning methods in seminar preparation and that the researchers would not intervene in the techniques they would create.
  Four different seminar groups were formed. There are 5 students in each group. Each group prepares a seminar on disaster nursing and management by using peer and self-learning methods.
  There are 20 students in this group. For 4 weeks, the groups made seminar presentations for 150 minutes one day a week.
  All seminar groups came together in the last week and formed a group discussion on disaster nursing research and development activities.
  Interventions: Other: Peer and Self-Learning Group
- Control Group (No Intervention): It consists of students who are not included in the intervention groups. The control group continues the education process in the routine education programme.
  This group consists of 24 students.

INTERVENTIONS:
Other: Model Based Training — experimental group
  Arms: Intervention Group 1
Other: Peer and Self-Learning Group — experimental group
  Arms: Intervention Group 2

SUMMARY:
This study was planned to evaluate the effect of two different learning methods on the perception of disaster preparedness and competences related to disaster management in nursing students.

DETAILED DESCRIPTION:
Disasters are an important public health problem due to their unpredictable duration, disruptions in society and health services, loss of life and property, significant economic losses, deterioration in psycho-social welfare and their effects in subsequent periods. Disaster events are events that exceed the local response capacity, where existing resources are insufficient in demand and require external assistance at international level. Therefore, disasters should be addressed not only in terms of their devastating effects but also in terms of the appropriate preparedness of the available resources in the community. Especially in the event of a disaster, it is certain that the demand for life-threatening medical care will increase, and the presence of timely accessible, equipped and prepared health workers is very important in disaster response.

Considering the increasing frequency of disasters and large-scale public health emergencies, this situation makes the disaster-related aspects of nursing particularly important. Nurses can serve as first responders, direct health care providers, point of care coordinators, information sources, educators and counsellors in disaster areas. However, most nurses and nursing students are not properly prepared for disaster situations.

Many disaster nursing education programmes are offered as themes within existing courses (health protection and promotion, public health and emergency nursing courses) through elective courses, seminars and conferences. As in many other areas of undergraduate nursing education, disaster education often adopts traditional instructor-centred teaching methods. According to the students' point of view, this teaching strategy has a monotonous and boring structure and may negatively affect the students' willingness to learn by shortening their attention span.

Simulation and scenario-based disaster nursing education programmes using standardised patients can be useful in disaster nursing education by improving students' skills and preparation. In case of disaster, models allow nurses to provide better service and performance.

In addition, peer-assisted and self-directed learning method content and teaching strategies aim to improve students' autonomy by incorporating students' feedback and comments into the design of the course. Student-centred education can consist of a variety of teaching tools and techniques, online audio-visual materials, activities, games and storytelling that reflect students' preferences. The student-centred education approach plays an important role in supporting the public health infrastructure and is receiving increasing attention in studies related to disaster preparedness and response.

In this study, it is aimed to evaluate the effect of two different learning methods on the perception of disaster preparedness and competencies related to disaster management in nursing students.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older Active student registration in the system between the specified dates Accepted to participate in the study verbally and in writing after being informed Who have not received training on disaster management before General health status (systemic, consciousness, sensation) is suitable for the research process

Exclusion Criteria:

* Having theoretical/practical training on disaster management Non-volunteering

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Introductory information form | All groups were administered a pre-test before the intervention, a post-test at the end of the 5-week intervention, a 1-month follow-up, a 3-month follow-up and a 6-month follow-up.
  The form, which was created by the researchers within the scope of the literature, includes 12 questions including socio-demographic characteristics, disaster experience, experience, and disaster-related information sources.
Nurses' Perception of Disaster Preparedness Scale | Pre-test before intervention, post-test at the end of 5-week intervention, 1-month follow-up, 3-month follow-up and 6-month follow-up stages were applied to all groups.
  This scale was developed by Feride Özcan in 2013 to measure how prepared nurses feel themselves against disasters. The scale consists of 20 items and 3 sub-dimensions as Preparation Phase (Questions 1-6), Intervention Phase (Questions 7-15), Post-Disaster Phase (Questions 16-20). The items of the scale are scored in five-point Likert type (1-Strongly disagree, 2-Disagree, 3-Somewhat agree, 4-Agree, 5-Strongly agree). As the score obtained from the scale increases, the perception of disaster preparedness also increases.

SECONDARY OUTCOMES:
Nurses' Competence Assessment Scale for Disaster Management | Pre-test before intervention, post-test at the end of 5-week intervention, 1-month follow-up, 3-month follow-up and 6-month follow-up stages were applied to all groups.
  The scale developed by Yıldız Keskin (2023) to evaluate the competences of nurses regarding disaster management consists of 43 items in two dimensions (disaster preparedness and disaster response). The items of the scale are scored in five-point Likert type (1-Strongly disagree, 2-Disagree, 3-Somewhat agree, 4-Agree, 5-Strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I want to share my research protocol after one year.

REFERENCES:
- See also: Related Info — https://www.who.int/activities/implementing-health-emergency-and-disaster-risk-management